CLINICAL TRIAL: NCT03207022
Title: Comparison Between Epinephrine and Clonidine as Adjuvants to Lidocaine in Ultrasound Guided Axillary Brachial Plexus Block.
Brief Title: Comparison Between Epinephrine and Clonidine as Adjuvants to Lidocaine in Axillary Brachial Plexus Block.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cork University Hospital (Other)
Responsible Party: Principal Investigator, Dr Anil Ranganath, Dr (Fellow in Regional Anaesthesia), Cork University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ECM 4 (aa)
Record Dates: First submitted 2017-05-07; First posted 2017-07-02 (Actual); Results first posted 2021-09-02 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Brachial Plexus Blockade

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lidocaine 2% with normal saline (Active Comparator): Patients will receive ultrasound guided axillary brachial plexus block with 20 ml of lidocaine 2% with epinephrine mixed with 2 ml of 0.9% normal saline.
  Interventions: Procedure: axillary brachial plexus block
- lidocaine 2% with clonidine (Experimental): Patients will receive ultrasound guided axillary brachial plexus block with 20 ml of lidocaine 2% with epinephrine mixed with clonidine 1µg/kg in 2 ml of 0.9% normal saline.
  Interventions: Procedure: axillary brachial plexus block

INTERVENTIONS:
Procedure: axillary brachial plexus block — ultrasound guided axillary brachial plexus block with 20 ml local anaesthetic lidocaine with epinephrine and clonidine

SUMMARY:
Adjuncts to local anaesthetics for the peripheral nerve blocks such as epinephrine, clonidine and opioids have been widely used to enhance quality, duration of anaesthesia and postoperative analgesia. Clonidine, an α2-adrenergic agonist, when combined with local anaesthetics in axillary brachial plexus block has shown to decrease block onset time and prolong the duration of anaesthesia.

We propose to compare the effects of combining both adjuvants to 20 mL of lidocaine 2% on the onset of ultrasound guided axillary brachial plexus block.

DETAILED DESCRIPTION:
Using a 20 mL lidocaine 2% when combined with epinephrine 1:200 000 and clonidine 1 µg/kg will shorten the onset time of sensory block when compared to lidocaine 2% with epinephrine 1:200 000 alone in ultrasound guided axillary brachial plexus block for elective upper limb surgeries.

It is a prospective, randomized, observer blinded study. With institutional ethical approval and having obtained written informed consent from each, 24 patients will be studied.

Randomisation and blinding:

Using a computer generated and sealed envelope technique, 24 patients will be randomized in to one of two groups to receive ultrasound guided axillary brachial plexus block.

Group 1:

Patients will receive 20 ml of lidocaine 2% with epinephrine and 2 ml of 0.9% normal saline.

Group 2:

Patients will receive 20 ml of lidocaine 2% with epinephrine and clonidine 1µg/kg in 2 ml of 0.9% normal saline.

Sample size and Statistical analysis:

Sample size will be based on onset of block. Kaabachi et al16 found a sensory onset of axillary brachial plexus block (with 30 ml of lidocaine 1.5%) of 9 (SD, 3) mins. The sample size required to have an 90% probability of detecting a decrease in the onset time by 40% (level of significance 0.05)) will be 12 patients per group using an unpaired student's t test.

Anaesthetic procedure:

Having established intravenous access, standard anaesthetic monitoring will be applied. Sedation with midazolam will be administered as clinically indicated (to a maximum of 3 mg). The operative arm will be abducted and externally rotated with elbow flexed at 90 degrees. Under strict aseptic condition, ultrasound guided axillary brachial plexus block will be performed. Having identified musculocutaneous, median, radial and ulnar nerves, a 50mm 22-gauge ultrauplex short bevel insulated needle will be used with in-plane approach to block each nerve. 20 mL of Lidocaine 2% with epinephrine and 2ml of 0.9% Nacl(group 1) or clonidine 1µg/kg in 2 ml of 0.9% Nacl(group 2) will be divided equally among the 4 nerves. All blocks will be performed by single operator experienced in the ultrasound peripheral nerve blocks.

Block assessment:

When the block procedure has been completed, a blinded observer will assess the onset of sensory and motor block in the innervation of each nerve every 2.5 mins until complete sensory and motor block is achieved or 30 mins have elapsed . Complete sensory block is defined as absent sensation to cold and pinprick and complete motor block is defined as motor score ≤2. Each nerve distribution will be individually assessed. Onset time will be measured from conclusion of the block (t=0) to attainment of (surgical anaesthesia) complete sensory and motor block. Block will be deemed failure if sensory and motor block has not been achieved at 30 mins in one or more of the four nerve distribution. In case of failure, an additional rescue block or conversion to general anaesthesia will be performed. DATA from these patients will be analysed separately.

Intraoperative period:

All patients will receive 1 g of paracetamol and diclofenac 75 mg iv during surgery. In case of patients discomfort rescue analgesia in the form of fentanyl 25 micrograms aliquots IV will be administered to a maximum of 100 micrograms.

Postoperative period:

Upon arrival to recovery room, sensory and motor function will be assessed every 15 mins by a blinded observer. Assessment will be performed for each nerve separately. Block regression is defined as a return of sensation to cold and pinprick with motor power score ≥3 in any nerve region. Time to first request for postoperative analgesia will be noted. Postoperative analgesia will be prescribed as paracetamol 1 g 6 hourly and diclofenac sodium 75 mg 12 hourly. Oxycodone 5-10 mg orally 4-6 hourly will be administered as rescue analgesia.

Heart rate, arterial blood pressure, spo2 and sedation score (1=awake and alert, 2= sedated, responding to verbal stimulus, 3= sedated, responding to mild physical stimulus and 4=sedated, responding to moderate to severe physical stimulus) will be recorded intraoperatively every 5 mins and every 15 mins postoperatively for the first 4 hours. Hypotension and bradycardia, defined as 20% decrease in blood pressure and heart rate in relation to preblock value, will be recorded.

Primary Outcome:

The primary outcome will be onset of sensory block.

Secondary Outcomes:

1. Onset of motor block.
2. Duration of sensory and motor block
3. The quality of block intra operatively
4. The incidence of side effects in both groups. : sedation, hypotension, nausea, dizziness, tinnitus, vomiting convulsions or arrthymia

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-2
* Patients age >18 years
* Undergoing elective upper limb (forearm, wrist or hand) surgery.

Exclusion Criteria:

* Contraindications to regional anaesthesia
* Hypersensitivity to amide local anaesthetics.
* Chronic pain
* Language barrier
* Neuromuscular disorders or peripheral neuropathy
* H/o postural hypotension or autonomic dysfunction.
* Patients with a known sensitivity for local anaesthetics
* Body mass index > 35
* History of hepatic and renal insufficiency
* Pregnancy
* Cognitive or psychiatric disorder
* Cardiac conduction abnormality.
* Anti arrythmic or adrenergic medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-06-11 (Actual); Primary Completion 2016-07-14 (Actual); Study Completion 2016-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anil Ranganath, Principal Investigator — Cork University Hospital

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Assessed for eligibility: n = 50 Excluded 26
  * Not meeting inclusion criteria n= 8
  * Declined to participate n= 18 Randomized n = 24
Period: Overall Study
Arm/Group | Lidocaine 2% With Normal Saline | Lidocaine 2% With Clonidine
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lidocaine 2% With Normal Saline | Lidocaine 2% With Clonidine | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.4 (10.6) | 42.3 (8.6) | 41.9 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 7 | 8 | 15
Region of Enrollment [Count of Participants; unit: Participants]
  Ireland | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Onset of Sensory Block
Description: Time taken for onset of sensory axillary brachial plexus block
Time Frame: 1 day
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Lidocaine 2% With Normal Saline | Lidocaine 2% With Clonidine
Number analyzed (Participants) | 12 | 12
minutes | 10 [8.8 to 12.5] | 5 [5 to 7.5]
Statistical Analysis 1: Comparison: Lidocaine 2% With Normal Saline vs Lidocaine 2% With Clonidine; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Onset of Motor Block.
Description: time taken for onset of motor block of ultrasound guided axillary brachial plexus block
Time Frame: 1 day
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Lidocaine 2% With Normal Saline | Lidocaine 2% With Clonidine
Number analyzed (Participants) | 12 | 12
minutes | 7.5 [6.3 to 7.5] | 5 [2.5 to 7.5]
Statistical Analysis 1: Comparison: Lidocaine 2% With Normal Saline vs Lidocaine 2% With Clonidine; Test type: Other; p = 0.001, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Duration of Sensory and Motor Block
Description: Total duration of sensory block of ultrasound guided axillary brachial plexus block
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Lidocaine 2% With Normal Saline | Lidocaine 2% With Clonidine
Number analyzed (Participants) | 12 | 12
minutes | 165 (24.1) | 218.3 (28.5)
Statistical Analysis 1: Comparison: Lidocaine 2% With Normal Saline vs Lidocaine 2% With Clonidine; Test type: Other; p < 0.001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 1 DAY
Description: The incidence of side effects in both groups. : sedation, hypotension, nausea, us, vomiting convulsions or arrythmia
Arm/Group | Lidocaine 2% With Normal Saline | Lidocaine 2% With Clonidine
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No